CLINICAL TRIAL: NCT07120711
Title: Regulatory Mechanisms of EGR2 and NLRP3 Inflammatory Pathways in Cognitive Impairment and Depressive-Anxiety-Like Behaviors Associated With Obstructive Sleep Apnea-Hypopnea Syndrome
Brief Title: EGR2 and NLRP3 Pathways in Obstructive Sleep Apnea-Related Cognitive and Mood Disorders
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai Jiang, 021-25077820, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2025-163-1
Record Dates: First submitted 2025-08-07; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea-Hypopnea Syndrome; Anxiety Disorders; Depressive Disorders
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- OSAS_chlidren
  Interventions: Procedure: EGR2/NLRP3 pathway activity
- OSAS_adult
  Interventions: Procedure: EGR2/NLRP3 pathway activity; Procedure: fatty tissue
- non_OSAS_chlidren
  Interventions: Procedure: EGR2/NLRP3 pathway activity
- non_OSAS_adult
  Interventions: Procedure: EGR2/NLRP3 pathway activity; Procedure: fatty tissue

INTERVENTIONS:
Procedure: EGR2/NLRP3 pathway activity — Peripheral blood collection & PBMC isolation:
  Children: 3 mL venous blood drawn from the right antecubital vein preoperatively; Adults: 3 mL fasting venous blood drawn the morning after PSG.
  Collected in EDTA tubes; PBMCs separated via Ficoll-Paque density gradient. Flow cytometry: 1×10⁶ PBMCs stained for CD14/CD16, HLA-DR, CD11b, CD80/CD86, CD163/CD206.
  RNA extraction: Remaining PBMCs lysed in TRIzol and stored at -80 °C for RT-qPCR of EGR2, NLRP3, and downstream genes Serum/plasma: Within 1 h of collection, centrifuge at 400 × g for 10 min at 4 °C; 1 mL used for ELISA quantification of TNF-α, IL-6, IL-1β, CCL2, IL-17, CRP; remainder stored at -80 °C for future proteomic or metabolomic assays
  Saliva sampling & processing:
  2-3 mL unstimulated saliva expectorated into sterile tubes, kept at 4 °C, processed (centrifuged, aliquoted) within 2 h, then stored at -80 °C.
Procedure: fatty tissue — Subcutaneous fat biopsy (adults undergoing surgery):
  100-200 mg obtained intraoperatively, placed in RNAlater at 4 °C for 24 h, then frozen at -80 °C for downstream RNA-seq, RT-qPCR, and Western blot analyses of EGR2, NLRP3, and related inflammatory markers
  Groups: OSAS_adult; non_OSAS_adult

SUMMARY:
Obstructive sleep apnea-hypopnea syndrome (OSAS) is a common disorder in which repeated airway blockages during sleep lead to low oxygen levels, inflammation, and disrupted sleep. Many OSAS patients-both children and adults-experience problems with memory, attention, and mood, such as anxiety or depression. However, the exact molecular drivers of these brain changes are not fully understood.

This observational study will enroll:

Children (ages 2-18) and adults (>18 years) with OSAS, as well as age- and sex-matched healthy volunteers.

Clinical assessments: Children will undergo routine ENT examinations (including nasal endoscopy and X-rays); adults will have an overnight sleep study (polysomnography). All participants will complete questionnaires on sleepiness (e.g., ESS), mood (PHQ-9, GAD-7), and cognitive screening (MoCA for adults, age-appropriate scales for children).

Sample collection: A small blood draw (3 mL) and, when applicable (e.g., adults undergoing surgery), a tiny subcutaneous fat biopsy. Saliva samples will also be collected.

Laboratory tests:

Measure expression levels of two key inflammatory pathway genes-EGR2 and NLRP3-in blood cells, saliva, and fat tissue using RNA sequencing, RT-qPCR, and Western Blot.

Correlate these molecular markers with sleep parameters (AHI, oximetry), cognitive scores, and mood scores.

Data analysis: Develop and validate machine-learning models that integrate data from multiple tissues to predict who is at highest risk for cognitive or mood disturbances.

ELIGIBILITY:
Inclusion Criteria:

Children aged 2-18 years with obstructive snoring or sleep apnea features on initial ENT outpatient screening.

Adults (>18 years) with suspected OSAS in a sleep or respiratory clinic, presenting with chronic snoring, witnessed apneas, or daytime sleepiness, and without severe chronic heart, liver, kidney failure, psychiatric disorders, or pregnancy.

Signed written informed consent by the participant or their legal guardian. Not currently enrolled in any other registered clinical trial.

Exclusion Criteria:

Presence of congenital craniofacial malformations. Severe heart, lung, liver, or kidney failure, or major neurological disease. Recent use of anti-inflammatory or other immunomodulatory medications. Current psychiatric disorder or pregnancy

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: his observational study will enroll both pediatric and adult participants with obstructive sleep apnea-hypopnea syndrome (OSAS) alongside age-matched healthy controls. Specifically:
  Pediatric cohort (2-18 years): Four age strata (2-6, 7-9, 10-12, 13-18 years), each with 50 OSAS patients and 50 healthy controls.
  Adult cohort (>18 years): Four age strata (18-40, 41-60, 61-80, >80 years), each with 50 OSAS patients and 50 healthy controls.
  Participants will be recruited from the ENT outpatient and sleep/respiratory clinics of Shanghai Xinhua Hospital and the MED-X Research Institute, Shanghai Jiao Tong University, between July 2025 and September 2026.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Expression levels of EGR2 and NLRP3 in PBMCs, saliva, and subcutaneous fat tissue | Jul 2025 - Sep 2026
  Quantitative measurement of EGR2 and NLRP3 mRNA (by RNA-seq and RT-qPCR) and protein levels (by Western blot and ELISA) in peripheral blood mononuclear cells, saliva, and (when available) subcutaneous fat tissue collected at baseline. These molecular markers will be correlated with cognitive (MoCA) and mood (PHQ-9, GAD-7) scores

SECONDARY OUTCOMES:
Multi-omics association of molecular markers with clinical phenotypes | Jul 2025 - Sep 2026
  Integration of transcriptomic (RNA-seq) and proteomic/metabolomic data from PBMC, saliva, and fat samples. Construction of weighted gene co-expression network analysis (WGCNA) modules and core protein-protein interaction (PPI) networks centered on EGR2/NLRP3, with annotation of inflammation and blood-brain barrier pathways; assessment of module eigengene correlations with AHI, minimum SpO₂, MoCA, PHQ-9, and GAD-7 scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xinhua hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No